CLINICAL TRIAL: NCT05759897
Title: A 16-week Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of HRS-7535 in Adults With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Brief Title: A 16 Week Study of HRS-7535 in Adults With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HRS-7535-201
Record Dates: First submitted 2023-02-09; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: HRS-7535 tablet compared with placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): Subjects will receive HRS-7535 administered orally
  Interventions: Drug: HRS-7535
- Group B (Experimental): Subjects will receive HRS-7535 administered orally
  Interventions: Drug: HRS-7535
- Group C (Experimental): Subjects will receive escalated dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535
- Group D (Experimental): Subjects will receive escalated HRS-7535 administered orally
  Interventions: Drug: HRS-7535
- Group E (Placebo Comparator): Subjects will receive Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-7535 — HRS-7535
  Arms: Group A; Group B; Group C; Group D
Drug: Placebo — Placebo
  Arms: Group E

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of HRS-7535 in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 age years, both inclusive;
2. Type 2 diabetes mellitus diagnosed for at least 3 months before the screening visit;
3. HbA1c 7.5-11.0% (both inclusive) by local laboratory analysis;
4. Treated with conventional lifestyle intervention and stable treatment with metformin (≥1000 mg/day) at least 8 weeks prior to screening.
5. Body weight of at least 50 kg; and Body Mass Index (BMI) within the range of 19 to 40 kg/m2 (inclusive);

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug or its components or excipients.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. Have a history of acute complications of diabetes (diabetic ketoacidosis, lactic acidosis, hyperglycaemic hyperosmolar state, etc.) within 6 months prior to screening.
4. Proliferative retinopathy, maculopathy, painful diabetic neuropathy, diabetic foot ulcer or intermittent claudication requiring acute treatment;
5. History or presence of vital organ primary diseases, including but not limited to neuropsychiatric, cardiovascular, digestive, respiratory, urinary, endocrine, blood, immune and other diseases, judged by researchers to be unsuitable for this study.
6. Discontinuation of previous glucagon-like peptide-1 receptor agonist therapy due to safety/tolerability reasons or lack of efficacy reasons.
7. Previous history of significant gastrointestinal disease (e.g. gastroesophageal reflux, gastric outlet obstruction, inflammatory bowel disease, active ulcers, etc.), or previous gastrointestinal surgery (except gastrointestinal polypectomy and appendectomy).
8. Pregnancy, breast-feeding, intention of becoming pregnant during the trial; or women of childbearing potential (WOCBP) or male subject not using adequate contraceptive measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-12-21 (Estimated); Study Completion 2024-01-04 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in HbA1c at Week 16 | at Week 16]

SECONDARY OUTCOMES:
Proportion of subjects reaching HbA1c targets (<7.0%) at Week 16 | at Week 16
Change From Baseline in fasting plasma glucose (FPG) at Week 16 | at Week 16
Change From Baseline in Mixed meal test at Week 16 | at Week 16
Change From Baseline in body weight at Week 16 | at Week 16
Change From Baseline in waist circumference at Week 16 | at Week 16
Change From Baseline in 7-point SMBG at Week 16 | at Week 16
Proportion of subjects receiving glycemic rescue medicine at Week 16 | at Week 16
A summary of adverse events, including serious adverse events (SAEs), and Hypoglycemic Event[ | at Week 18

IPD SHARING:
Plan to Share IPD: Undecided